CLINICAL TRIAL: NCT01717209
Title: Combined Inhaled Nitric Oxide and Inhaled Prostacyclin After Cardiac Surgery for Heart Transplantation and for Left Ventricular Assist Device Placement
Brief Title: Inhaled Nitric Oxide and Inhaled Prostacyclin After Cardiac Surgery for Heart Transplant or LVAD Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Charles Hill, Clinical Associate Professor, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25471
Record Dates: First submitted 2012-10-26; First posted 2012-10-30 (Estimated); Results first posted 2017-10-09 (Actual); Last update posted 2017-10-09 (Actual); Status verified 2017-10

CONDITIONS: Heart Failure
Keywords: heart failure; hypertension, pulmonary; heart failure, right-sided; heart-assist devices; Heart Transplantation
MeSH Terms: conditions — Heart Failure; Hypertension, Pulmonary | interventions — Nitric Oxide; Endothelium-Dependent Relaxing Factors; Epoprostenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Combined nitric oxide and prostacyclin (Experimental): iNO (20 ppm continuously) and iPGI2 (0.05 micrograms/kg/min continuously)
  Interventions: Drug: Nitric Oxide; Drug: Prostacyclin

INTERVENTIONS:
Drug: Nitric Oxide — inhaled nitric oxide
  Other Names: INOmax
Drug: Prostacyclin — inhaled prostacyclin
  Other Names: inhaled flolan; epoprostenol; inhaled PGI2

SUMMARY:
Research study evaluating the individual and combined effects of inhaled nitric oxide (iNO) and inhaled prostacyclin (iPGI2), on the function of the right heart after surgery for either heart transplant or for left ventricular assist device (LVAD) placement. The investigators hope to learn if these two medications, when given together after surgery, improve right heart function by lowering blood vessel pressures in the lungs. The investigators hope to learn if the combined effects of these two medications are better than either medication used alone. Participants were selected as a possible participant in this study because right heart problems are common during and after surgery for heart transplant and for LVAD placement. In addition, iNO is always given during and after these two types of surgeries at Stanford to help improve how the right heart functions.

DETAILED DESCRIPTION:
The study will begin once the participant arrives in the cardiothoracic intensive care unit (CTICU) after heart surgery for either heart transplant or LVAD placement. As is standard of care after these types of surgeries, the participant will arrive in the CTICU with a breathing tube already in place, receiving iNO, and connected to a breathing machine. The participant will be receiving relaxing medication in an intravenous line provided by the cardiac anesthesiologist and the CTICU physicians. The participant will be unaware of the study period while the participant is sedated. Data will be collected from the monitor screen connected to the participant's arterial and venous lines, and if placed, LVAD monitor. These data are:

Central venous pressure (CVP) Mean arterial pressure (MAP) Mean pulmonary artery pressure (MPAP) Cardiac Index (CI) Systemic vascular resistance (SVR) Pulmonary vascular resistance (PVR) Right ventricular stroke work index (RVSWI) LVAD Flow LVAD Pulsatility Index (PI)

These data will be collected at five different time periods during the first eight hours after surgery.

1. Time zero. Data will be collected after surgery upon your arrival to the CTICU while receiving iNO.
2. After two hours of iNO treatment data will be collected. iPGI2 will then be combined with the current iNO.
3. After two hours of combined iNO and iPGI2 treatment, data will be collected. iNO will then be stopped.
4. After two hours of iPGI2 treatment data will be collected. iNO will be restarted.
5. After two hours of combined iNO and iPGI2 treatment, data will be collected. The study ends after this data collection time.

ELIGIBILITY:
Inclusion Criteria:

* Adult cardiac surgical patients scheduled to undergo either heart transplantation or LVAD placement

Exclusion Criteria:

* Patients with prior documented allergic reactions or intolerance to either nitric oxide or prostacyclin will be excluded. Patients not undergoing heart transplantation or LVAD placement will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10 (Actual); Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew J Powers, MD, Principal Investigator
Locations (1):
- Stanford Hospital and Clinics, Stanford, California, United States

REFERENCES:
- [Background] Khan TA, Schnickel G, Ross D, Bastani S, Laks H, Esmailian F, Marelli D, Beygui R, Shemin R, Watson L, Vartapetian I, Ardehali A. A prospective, randomized, crossover pilot study of inhaled nitric oxide versus inhaled prostacyclin in heart transplant and lung transplant recipients. J Thorac Cardiovasc Surg. 2009 Dec;138(6):1417-24. doi: 10.1016/j.jtcvs.2009.04.063. PMID 19931670
- [Background] De Wet CJ, Affleck DG, Jacobsohn E, Avidan MS, Tymkew H, Hill LL, Zanaboni PB, Moazami N, Smith JR. Inhaled prostacyclin is safe, effective, and affordable in patients with pulmonary hypertension, right heart dysfunction, and refractory hypoxemia after cardiothoracic surgery. J Thorac Cardiovasc Surg. 2004 Apr;127(4):1058-67. doi: 10.1016/j.jtcvs.2003.11.035. PMID 15052203
- [Background] Potapov E, Meyer D, Swaminathan M, Ramsay M, El Banayosy A, Diehl C, Veynovich B, Gregoric ID, Kukucka M, Gromann TW, Marczin N, Chittuluru K, Baldassarre JS, Zucker MJ, Hetzer R. Inhaled nitric oxide after left ventricular assist device implantation: a prospective, randomized, double-blind, multicenter, placebo-controlled trial. J Heart Lung Transplant. 2011 Aug;30(8):870-8. doi: 10.1016/j.healun.2011.03.005. Epub 2011 Apr 29. PMID 21530317
- [Background] Antoniou T, Prokakis C, Athanasopoulos G, Thanopoulos A, Rellia P, Zarkalis D, Kogerakis N, Koletsis EN, Bairaktaris A. Inhaled nitric oxide plus iloprost in the setting of post-left assist device right heart dysfunction. Ann Thorac Surg. 2012 Sep;94(3):792-8. doi: 10.1016/j.athoracsur.2012.04.046. Epub 2012 Jun 23. PMID 22727248

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined Nitric Oxide and Prostacyclin: Inhaled nitric oxide (iNO; 20 ppm continuously) and inhaled prostacyclin (iPGI2; 0.05 micrograms/kg/min continuously)
Period: Overall Study
Arm/Group | Combined Nitric Oxide and Prostacyclin
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
Age, Continuous [Mean (Full Range); unit: years] | 57 [29 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Pulmonary Hypertension
Description: Pulmonary hypertension was measured as mean of Mean Pulmonary Artery Pressure for initial 8 hours after admission to the Intensive Care Unit (ICU). MPAP value ≥25 mmHg (resting) indicates pulmonary hypertension state.
Time Frame: 8 hours (upon arrival at ICU, and after 4 successive 2 hour treatments with 1. iNO only, 2. iNO+iPGI2 (1st), 3. iPGI2 only, and 4. iNO+iPGI2 (2nd))
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
mmHg
  At Arrival in ICU | 31.4 [20 to 43]
  Following iNO | 29.1 [16 to 44]
  Following iNO+iPGI2 (1st) | 25.9 [17 to 36]
  Following iPGI2 | 25.4 [15 to 38]
  Following iNO+iPGI2 (2nd) | 25.4 [12 to 46]

2. Secondary Outcome: Right Heart Dysfunction
Description: Right Heart Dysfunction was measured as mean of Right Ventricular Stroke Work Index (RVSWI) for the initial 8 hours after admission to the Intensive Care Unit (ICU). RVSWI is measured as the difference in mean pulmonary artery pressure (MPAP) and central venous pressure (CVP), divided by the cardiac index (CI): [(MPAP-CVP) / CI]. Normal range for RVSWI is 5-10 g/m.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: g/m
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
g/m
  At Arrival in ICU | 5.2 [2.64 to 11.15]
  Following iNO | 5.0 [1.45 to 9.06]
  Following iNO+iPGI2 (1st) | 4.8 [1.96 to 8.40]
  Following iPGI2 | 5.4 [2.10 to 13.14]
  Following iNO+iPGI2 (2nd) | 4.9 [1.30 to 10.05]

3. Secondary Outcome: Systemic Vascular Resistance (SVR)
Description: Systemic Vascular Resistance (SVR) was measured as mean of Systemic Vascular Resistance (SVR) for the initial 8 hours after admission to the Intensive Care Unit (ICU). Normal range for SVR is 800-1200 dynes/sec/cm5.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: dynes/sec/cm^5
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
dynes/sec/cm^5
  At Arrival in ICU | 1193.9 [488.0 to 1542]
  Following iNO | 1169.7 [898.0 to 1945]
  Following iNO+iPGI2 (1st) | 1070.6 [736.0 to 1520]
  Following iPGI2 | 1132.4 [711.00 to 1640]
  Following iNO+iPGI2 (2nd) | 1145.9 [783.0 to 1649]

4. Secondary Outcome: Central Venous Pressure (CVP)
Description: Central Venous Pressure (CVP) was measured as mean of CVP for the initial 8 hours after admission to the Intensive Care Unit (ICU). Normal range for CVP is 3-8 mmHg.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
mmHg
  At Arrival in ICU | 12.7 [4 to 19]
  Following iNO | 12.6 [5 to 18]
  Following iNO+iPGI2 (1st) | 11.6 [6 to 15]
  Following iPGI2 | 10.1 [2 to 15]
  Following iNO+iPGI2 (2nd) | 10.6 [4 to 14]

5. Secondary Outcome: Mean Arterial Pressure (MAP)
Description: Mean Arterial Pressure (MAP) was measured as mean of MAP for the initial 8 hours after admission to the Intensive Care Unit (ICU). Normal range for MAP is 70-110 mmHg.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: mmHg
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
mmHg
  At Arrival in ICU | 86.29 [68 to 102]
  Following iNO | 80.86 [62 to 91]
  Following iNO+iPGI2 (1st) | 79.00 [67 to 89]
  Following iPGI2 | 79.43 [63 to 91]
  Following iNO+iPGI2 (2nd) | 80.86 [61 to 103]

6. Secondary Outcome: Heart Rate
Description: Heart Rate was measured as mean of Heart Rate for the initial 8 hours after admission to the Intensive Care Unit (ICU). Normal range for heart rate is generally 60 to 100 beats per minutes in adults, but this can vary.
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: beats/minute
Arm/Group | Combined Nitric Oxide and Prostacyclin
Number analyzed (Participants) | 14
beats/minute
  At Arrival in ICU | 111.1 [75 to 152]
  Following iNO | 112.5 [71 to 166]
  Following iNO+iPGI2 (1st) | 108.4 [73 to 161]
  Following iPGI2 | 106.0 [67 to 134]
  Following iNO+iPGI2 (2nd) | 104.6 [73 to 119]

ADVERSE EVENTS:
Arm/Group | Combined Nitric Oxide and Prostacyclin
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

LIMITATIONS AND CAVEATS:
Analyses are underpowered due low enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No